CLINICAL TRIAL: NCT05511896
Title: Effects of Repeated Trunk Flexion on Trunk Neuromuscular Properties.
Brief Title: Effects of a 60-min Repeated Trunk Flexion Protocol on Trunk Neuromuscular Properties.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Primorska (Other)
Responsible Party: Principal Investigator, MatejVoglar, Assistant professor, PhD, University of Primorska
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: SWE_Flexion1
Record Dates: First submitted 2022-08-19; First posted 2022-08-23 (Actual); Last update posted 2022-10-19 (Actual); Status verified 2022-10

CONDITIONS: Occupational Exposure
Keywords: bending, load, stiffness, elastography, deformation
MeSH Terms: conditions — Airway Obstruction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intermittent trunk flexion (Experimental): 60-min intermittent trunk flexion protocol.
  Interventions: Other: Repeated trunk flexion

INTERVENTIONS:
Other: Repeated trunk flexion — A 60-min intermittent trunk flexion protocol. Participants will sit on a standard height sit, with their knees bent at approximately 90° with their hands crossed on their chest. They will perform 40 sets of 60 s of maintaining a flexed position, interspersed with 30 s of rest. Participants will achieve the flexed position by tilting the pelvis posteriorly and leaning forward. During rest, participants will sit up straight without leaning on the support.

SUMMARY:
An interventional study on the effects of repeated trunk flexion exposure on trunk neuromuscular properties.

DETAILED DESCRIPTION:
An interventional study will include 16 healthy young adults. All participants will complete a 60-min protocol of intermittent trunk flexion. Measurements of trunk neuromuscular properties will be performed prior to and following the 60-min protocol.

ELIGIBILITY:
Inclusion Criteria:

* Physically active at least 3 hours a week

Exclusion Criteria:

* Low back pain in the past 6 months
* History of chronic low back pain
* History of spinal or pelvic operation
* Hypermobility, more than 4 points on Beighton scale
* Cardiovascular or systemic diseases
* Pregnancy

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2022-10-01 (Actual); Study Completion 2022-10-15 (Actual)

PRIMARY OUTCOMES:
Change in muscle stiffness | 90 minutes
  Muscle stiffness will be measured in prone lying using ultrasound-based shear wave elastography. Erector spinae and multifidus muscle stiffness will be expressed as the shear modulus value in kilopasquals.

SECONDARY OUTCOMES:
Change in range of motion | 90 minutes
  Trunk flexion range of motion will be evaluated using inertial measuring units during bending in standing position.
Change in length of the spine | 90 minutes
  The length of spine will be measured on a custom-developed stadiometer, with the participants in a seated position.
Change in muscle activity | 90 minutes
  Muscle activity will be measured using electromyography during standing.

CONTACTS AND LOCATIONS:
Overall Officials: Matej Voglar, PhD, Principal Investigator — University of Primorska, Faculty of Health Sciences
Locations (1):
- University of Primorska, Faculty of Health Sciences, Izola, Primorska, Slovenia

IPD SHARING:
Plan to Share IPD: Yes
Coded individual data will be uploaded on public scientific data repository.
Supporting Information: Study Protocol